CLINICAL TRIAL: NCT02545829
Title: A Randomized, Open, 2-way Cross-over, Single Dose Study to Evaluate and Compare Safety and Pharmacokinetics of the HIP1302 and HGP1406 (Tenofovir) in Healthy Korean Male Volunteers
Brief Title: Evaluating the Bioequivalence of HIP1302, HGP1406
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-POVI-101
Record Dates: First submitted 2015-08-13; First posted 2015-09-10 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): HGP1406 → HIP1302
  Interventions: Drug: HIP1302; Drug: HGP1406
- Sequence 2 (Experimental): HIP1302 → HGP1406
  Interventions: Drug: HIP1302; Drug: HGP1406

INTERVENTIONS:
Drug: HIP1302 — Tenofovir 292mg
Drug: HGP1406 — Tenofovir 300mg

SUMMARY:
The purpose of this study is to investigate the bioequivalence after administration of HIP1302 and HGP1406 in healthy male volunteers.

DETAILED DESCRIPTION:
A Randomized, Open, 2-way cross-over, Single dose study to Evaluate and Compare Safety and Pharmacokinetics of the HIP1302 and HGP1406 in Healthy Korean Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age 19 to 50 years
* The result of Body Mass Index(BMI) is not less than 18.0 kg/m2, no more than 27.0 kg/m2
* Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Tenofovir Cmax | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)
Tenofovir AUClast | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)

SECONDARY OUTCOMES:
Tenofovir Tmax | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)
Tenofovir t1/2 | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)
Tenofovir CL/F | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)
Tenofovir AUCinf | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)
Tenofovir MRT | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)
Tenofovir Vd/F | 0h(predose), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72hour (Total 16)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No